CLINICAL TRIAL: NCT03745807
Title: A Phase 1 Study to Evaluate Safety and Tolerability of NKTR-214 (BMS-986321) Administered in Combination With Nivolumab (BMS-936558) in Advanced Malignant Tumors
Brief Title: An Investigational Study of NKTR-214 Combined With Nivolumab in Japanese Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nektar Therapeutics (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA045-010; 18-214-14 (Other: Nektar Therapeutics)
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination (Experimental): NKTR-214 + nivolumab
  Interventions: Biological: NKTR-214; Biological: Nivolumab

INTERVENTIONS:
Biological: NKTR-214 — Specified dose on specified days
  Other Names: Bempegaldesleukin; BMS-986321
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to assess the safety and tolerability of NTKR-214 in combination with nivolumab in Japanese participants with advanced malignant tumors.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologic or cytological confirmation of an advanced (metastatic and/or unresectable) malignant solid tumor with measurable disease per RECIST v1.1.
* Life expectancy >12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Active, known or suspected autoimmune disease.
* History of organ transplant that requires use of immune suppressive agents.
* Prior surgery or radiotherapy within 14 days of Cycle 1 Day 1. Participants must have recovered from all radiation-related, toxicities and not requiring corticosteroids.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Approximately 2 years
Incidence of serious adverse events (SAEs) | Approximately 2 years
Incidence of AEs leading to discontinuation | Approximately 2 years
Incidence of deaths | Approximately 2 years
Incidence of AEs meeting protocol-defined dose limiting toxicity (DLT) criteria | Approximately 2 years
Incidence of laboratory abnormalities | Approximately 2 years

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Approximately 2 years
Time of maximum observed concentration (Tmax) | Approximately 2 years
Area under the concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Approximately 2 years
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Approximately 2 years
Total body clearance (CLT) | Approximately 2 years
Volume of distribution (Vz) | Approximately 2 years
Apparent terminal phase half-life (T-HALF) | Approximately 2 years
Trough observed serum concentration at the end of the dosing interval (Ctrough) | Approximately 2 years
Incidence of anti-drug antibodies (ADA) to NKTR-214 | Approximately 2 years
Incidence of anti-drug antibodies (ADA) to nivolumab | Approximately 2 years
Best overall response (BOR) | Approximately 2 years
Duration of response (DOR) | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data from this study may be shared with qualified researchers, upon request, following the timelines and process detailed on https://www.bms.com/researchers-and-partners/independent-research/data-sharing-request-process.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm